CLINICAL TRIAL: NCT06409741
Title: PrEveNtion of Biliary Events After Acute Pancreatitis in NonSUrgicaL PAtients. Sphincterotomy Vs Conservative Treatment. Multicenter Randomized Clinical Trial: PENINSULA Trial
Brief Title: PrEveNtion of Biliary Events After Acute Pancreatitis in NonSUrgicaL PAtients: PENINSULA Trial
Acronym: PENINSULA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario de Alicante (Other)
Collaborators: Hospital Universitario Ramon y Cajal (Other); Hospital del Rio Hortega (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government); Hospital Clínico Universitario de Valencia (Other)
Responsible Party: Principal Investigator, Jose Ramon Aparicio Tormo, Medical Doctor, Chief of Endoscopy Unit, Hospital General Universitario de Alicante
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEIm Ref: 2023-139 (2023-414)
Record Dates: First submitted 2024-05-05; First posted 2024-05-10 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Acute Pancreatitis Due to Gallstones; Acute Pancreatitis
Keywords: sphincterotomy; acute pancreatitis; recurrence; conservative treatment; biliopancreatic events
MeSH Terms: conditions — Pancreatitis; Recurrence | interventions — Sphincterotomy, Endoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biliary sphincterotomy (Active Comparator): In the group assigned to receive endoscopic treatment, ERCP for biliary sphincterotomy will be performed during the index admission for acute pancreatitis, prior to discharge or up till one month from discharge.
  The procedure will be performed after at least 6 hours of fasting during the index admission, by endoscopists in charge of performing ERCP as usual in the collaborating centers under sedation controlled by endoscopists or anesthesia according to the usual practice of the Endoscopy Unit of each collaborating center.
  For ERCP biliary cannulation, the usual techniques available in each center will be used, including advanced cannulation techniques if necessary.
  If biliary cannulation is not possible, a new ERCP attempt will be performed within a maximum of one month. If biliary cannulation is still not achieved, it will be counted as a technical failure.
  Interventions: Procedure: Biliary sphincterotomy
- Conservative treatment (No Intervention): Patients allocated to this group will be discharged without any intervention. The inhospital management of patients with AP in the conservative treatment group, before and after randomization, will be under the care of their responsible physicians on the hospitalization wart at the corresponding collaborating center who will follow the management recommended by the clinical guidelines. Their discharge will be decided by their regular physician. Patients will be evaluated at one month, six months and one year and both clinical variables (clinical BPE recurrence) and quality of life will be assessed (quality of life by a survey- EORTC QLQ-C30,

INTERVENTIONS:
Procedure: Biliary sphincterotomy — ERCP for biliary sphincterotomy will be performed during index admission for acute pancreatitis, prior to discharge or up till one month from discharge.
  The procedure will be performed after at least 6 hours of fasting during the index admission, by endoscopists in charge of performing ERCP as usual in the collaborating centers under sedation controlled by endoscopists or anesthesia according to the usual practice of the Endoscopy Unit of each collaborating center.
  For ERCP biliary cannulation, the usual techniques available in each center will be used, including advanced cannulation techniques if necessary.
  If biliary cannulation is not possible, a new ERCP attempt will be performed within a maximum of one month. If biliary cannulation is still not achieved, it will be it will be counted as a technical failure, maintaining the established clinical follow-up.
  Arms: Biliary sphincterotomy

SUMMARY:
Acute pancreatitis (AP) is a common condition and its main etiology is biliary. Cholecystectomy is the standard preventive treatment for recurrence of AP after admission. However, due to an increasingly older population and increased patient comorbidity, it is not always a possible option these days. If cholecystectomy is not performed, there is a significant risk for a recurrence of a biliopancreatic event (pancreatitis, biliary colic, choledocholithiasis, cholecystitis or cholangitis) of around 50% in the first year. This can lead to further episodes of pain, patient readmissions, and a reduced quality of life. Additionally, frequent readmissions can create a high cost burden on the health system. Currently, certain clinical guidelines propose biliary sphincterotomy as an alternative for patients in whom surgery is not feasible. However, this recommendation is based on retrospective studies with small sample size and the adherence to this recommendation is very low (12-23%).

The goal of this clinical trial is to evaluate the recurrence of biliopancreatic events in the first year after admission for an acute biliary pancreatitis episode in patients that are not suitable for surgery. The main question it aims to answer is:

Does biliary sphincterotomy prevent biliopancreatic event recurrence in non surgical patients after an episode of biliary acute pancreatitis?

Researchers will compare biliary sphincterotomy vs conservative treatment to see if there is a reduction in biliopancreatic events during the first year after admission for acute pancreatitis in non surgical patients.

Participants will be randomized to conservative treatment or biliary sphincterotomy and will be followed up for one year at 1 month, 6 months and 12 months to evaluate recurrence of BPE, readmissions, quality of life and mortality. Security of the technique will also be assessed in this specific population.

DETAILED DESCRIPTION:
Our working hypothesis is that endoscopic treatment with biliary sphincterotomy will reduce the number of biliopancreatic events compared to conservative treatment in patients with non-operable biliary acute pancreatitis (AP) due to a high surgical risk or in those patients who refuse surgery.

The primary aim is to assess the recurrence of the combined variable of biliopancreatic events (BPE) (biliary colic, cholangitis, choledocholithiasis, acute cholecystitis or AP) of the endoscopic sphincterotomy strategy during the follow-up time after diagnosis of AP of biliary origin in inoperable patients with respect to conservative treatment.

This is a randomized, multicenter, open-label, nationwide, intention-to-treat clinical trial. Patients will be randomized 1:1 to the two treatment groups stratified by center and AP severity.

Centers considered to participate as collaborators centers will need to have an endoscopy unit with ERCP availability that perform more than 150 ERCPs/year, and endoscopists trained in this technique. Patient inclusion and exclusion criteria is specified in a specific section of the protocol.

For the inclusion of patients, after diagnosis of biliary AP (BAP), and having ruled cholecystectomy as a possibility for the patient because of high surgical risk (after evaluation by surgery or anesthesia) or patient's refusal to undergo cholecystectomy, the absence of choledocholithiasis will be confirmed by MRCP or EUS.

If the patient fulfills these requirements, in addition to all the previous inclusion criteria and none of the exclusion criteria, and agrees to participate in the study and signs the informed consent the patient will be included and randomized.

This randomization will be carried out in each of the collaborating centers and the patient will be assigned to a treatment group following the random assignment method.

The randomization of patients to each of the treatment groups will be carried out centrally by the REDCap software; REDCap is a program that offers an online electronic data collection notebook. It will be stratified by center and by severity of BAP (mild, moderate or severe according to the Revised Atlanta Classification).

Patients will be randomized to receive ERCP biliary sphincterotomy or conservative management. 63 patients will be allocated to each group. An interim safety analysis is proposed, which will be evaluated by an independent committee of 3 persons, with experience in complications associated with ERCP and knowledge of biliopancreatic pathology, once 50% of the sample reaches 6 months of follow-up. In the event that in this first analysis the risks of treatment outweigh the benefits, according to the decision of the safety committee, the study could be stopped. Also, in the event that at this point there are statistically significant differences in favor of treatment by biliary sphincterotomy with respect to the primary outcome, recruitment can be stopped and the study stopped early.

In the group assigned to receive endoscopic treatment, ERCP for biliary sphincterotomy will be performed during the index admission for acute pancreatitis, prior to discharge or up till one month from discharge.

The procedure will be performed after at least 6 hours of fasting during the index admission, by endoscopists in charge of performing ERCP as usual in the collaborating centers under sedation controlled by endoscopists or anesthesia according to the usual practice of the Endoscopy Unit of each collaborating center.

For ERCP biliary cannulation, the usual techniques available in each center will be used, including advanced cannulation techniques if necessary. The type of papilla, cannulation attempts, time to biliary cannulation and the technique(s) used will be recorded. Possible adverse effects will be recorded. If biliary cannulation is not possible, a new ERCP attempt will be performed within a maximum of one month. If biliary cannulation is still not achieved, it will be counted as a technical failure, maintaining the established clinical follow-up.

The inhospital management of patients with AP in the conservative treatment group, before and after randomization, will be under the care of their responsible physicians on the hospitalization wart at the corresponding collaboration center who will follow the management recommended by the clinical guidelines. Their discharge will be decided by their regular physician.

Periodic follow-up contacts will be made: at one month, at 6 months and at one year. Contacts may be made by face-to-face or telematic visits after consultation with the patient, especially if the patient is institutionalized or has severe mobility problems.

In these contacts, the following will be performed:

* Record of complications associated with the treatment received and record of BPE developed since the last visit (especially the presence of biliary colic that did not require admission or evaluation in the emergency department). An interview will be conducted aimed at collecting the presence of BPE that did not require admission (such as biliary colic or related pain), recording the type and date of onset. The digital medical record will also be reviewed to record admissions and assessments by the emergency department related or unrelated to BPE and also to assess mortality.
* EORTQ30 quality of life questionnaire will be conducted in every visit.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years old.
* Definitive diagnosis of acute pancreatitis according to the presence of two out of three criteria from the Revised Atlanta Classification. At least 2 criteria: A) Typical pain, B) Amylase or lipase ≥x3 normal limit, C) Imaging evidence compatible with acute pancreatitis).
* Biliary etiology: (any imaging test that describes gallbladder lithiasis/microlithiasis or biliary sludge).
* Magnetic resonance cholangiography (MRCP) or endoscopic ultrasound (EUS) is required without evidence of choledocholithiasis.
* Surgical decision of inoperable patient (if meets one or more of the following criteria: age ≥ 80 years, American Society of Anesthesiology (ASA) III or more, Charlson Comorbidity Index > 5 and/or Karnofsky < 50 or patient's decision not to undergo surgery. Patient must have been evaluated by general surgery or anesthesia.
* Signature of the informed consent for the study

Exclusion Criteria:

* Patient refusal to participate in the study.
* Active ethylism greater than or equal to 5 drinking units per day in men and 3 in women or strong clinical suspicion of clinically significant ethylism that could be a cause of their AP.
* Hypertriglyceridemia greater than 400 mg/dl at admission or history of poorly controlled hypertriglyceridemia.
* Chronic pancreatitis: pancreatic calcifications in body or Wirsung on imaging or Wirsung ≥ 4 mm
* Biliary condition requiring sphincterotomy during index admission (cholangitis or symptomatic choledocholithiasis) or previous biliary sphincterotomy.
* Previous cholecystectomy
* Actual use of ursodeoxycholic acid
* Gastrointestinal tract anatomy altered by previous hepatobiliary or upper gastrointestinal surgery.
* Inability to tolerate endoscopy sedation, perforation of the digestive tract or other contraindication to endoscopy.
* Coagulopathy with uncorrectable International Normalized Ratio > 1.5 or uncorrectable thrombocytopenia < 50000/mm3.
* Other concomitant diagnoses on admission (liver abscesses, biliopancreatic neoplasia, acute cholecystitis).
* Hemodynamic instability.
* Baseline ECOG ≥4

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Biliopancreatic events (BPE) | From enrollment until 12 months after
  The primary aim is to assess the recurrence of the combined variable of biliopancreatic events (biliary colic, cholangitis, choledocholithiasis, acute cholecystitis or AP) of the endoscopic sphincterotomy strategy during the follow-up time after diagnosis of AP of biliary origin in inoperable patients with respect to conservative treatment.

SECONDARY OUTCOMES:
Time to recurrence of BPE | From enrollment until 12 months after
  Time in days to recurrence of biliopancreatic events between both groups
Recurrence of each of the variables that make up the combined variable BPE separately | From enrollment until 12 months after
  To assess the recurrence of each of the variables that make up the combined variable BPE separately and compare them between groups (AP, cholangitis, choledocholithiasis, cholecystitis, biliary colic).
Technical success of biliary sphincterotomy | From enrollment until one month after
  Technical success will be defined as the achievement of biliary sphincterotomy defined by the endoscopist performing the procedure.
Sphincterotomy related adverse events | From enrollment until one month after
  To describe the complications associated with sphincterotomy and the management of these adverse events of patients included in the study with the AGREE scale of endoscopic adverse events (Classification of Adverse events GastRointEstinal Endoscopy). This classification of adverse events ranges from 0 (no adverse events) until 5 (death) due to complications related to the procedure.
Emergency room visits (BPE related) | From enrollment until 12 months after
  Number of visits to the emergency room due to a BPE
Admission rate (BPE related) | From enrollment until 12 months after
  To evaluate differences between admission rate in hospital between both groups related to BPE
Admission rate (not BPE related) | From enrollment until 12 months after
  Number of admissions (not directly associated to BPE) in hospital and comparison between both groups
Emergency room visits (not BPE related) | From enrollment until 12 months after
  Number of emergency room visits that do not require admission and are not specifically related to BPE
Mortality at 30 days | From enrollment until one month after
  Mortality at 30 days and comparison between both groups
Hospital readmission at 30 days | From enrollment until one month after
  Hospital admission at day 30 due to EBP or not related to EBP and comparison between both groups
Mortality at one year | From enrollment until 12 months after
  Evaluation of mortality at one year and comparison between both groups
Index admission duration | From enrollment until one month after
  Days of index admission due to AP and comparison between both groups
Quality of life during follow-up | From enrollment until 12 months after
  Quality of life will be assessed at every visit (1 month, 6 months and 12 months) with EORTC ( European Organization for Research and Treatment of Cancer ) Quality of Life Questionnaire C-30 and groups will be compared.The questionnaire is structured in 5 functional scales (physical functioning, activities of daily living, emotional functioning, cognitive functioning and social functioning), 3 symptom scales (fatigue, pain and nausea, vomiting), 1 global health status scale and, finally, 6 independent items (dyspnea, insomnia, anorexia, constipation, diarrhea and economic impact). Values between 1 and 4 (1: not at all, 2: a little, 3: quite a lot, 4: a lot) are assigned according to the patient's responses to the item, only items 29 and 30 are evaluated with scores from 1 to 7 (1: very bad, 7: excellent). The scores obtained are standardized and a score between 0 and 100 is obtained.

CONTACTS AND LOCATIONS:
Overall Officials: José R Aparicio, MD, Principal Investigator — Hospital General Universitario Dr. Balmis
Locations (5):
- Spain (5):
  - Hospital General Universitario Dr. Balmis, Alicante, Alicante
  - Hospital Universitaria Reina Sofía, Córdoba, Cordoba
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Clinico Universitairo, Valencia, Valencia
  - Hospital Universitario Río Hortega, Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No